CLINICAL TRIAL: NCT00003175
Title: A Phase II Study of Continuous 5-Fluorouracil (5-FU) in Recurrent Locally Advanced or Metastatic Transitional Cell Carcinoma of the Urinary Tract
Brief Title: Fluorouracil in Treating Patients With Recurrent or Metastatic Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065985; MRC-BA10; EU-97029
Record Dates: First submitted 1999-11-01; First posted 2004-04-30 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2010-02

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: recurrent bladder cancer; transitional cell carcinoma of the bladder; recurrent urethral cancer; recurrent transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Fluorouracil

INTERVENTIONS:
Drug: fluorouracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of fluorouracil given as a continuous infusion in treating patients with recurrent or metastatic bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and toxic effects of continuous fluorouracil in patients with recurrent locally advanced or metastatic transitional cell urinary tract carcinoma. II. Determine the feasibility of this treatment in this patient population.

OUTLINE: Patients receive continuous intravenous fluorouracil by a Baxter Infusor for 24 weeks. Patients are evaluated for complete and partial response at 8, 16, and 24 weeks after the start of intravenous fluorouracil. Patients experiencing disease progression or unacceptable toxic effects are removed from the study. Patients are followed monthly for 6 months post treatment.

PROJECTED ACCRUAL: A maximum of 45 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent locally advanced or metastatic transitional cell urinary tract carcinoma that has been previously untreated with systemic chemotherapy Pelvic relapse after radiotherapy or surgery No relapse solely within a previously irradiated field Nodal or metastatic disease Lesions within the abdomen or pelvis must be assessed using CT scanning At least one site of disease must be previously unirradiated and assessable for response Bone metastases cannot be used as an indicator lesion Measurable disease

PATIENT CHARACTERISTICS: Age: Not specified Performance Status: Not specified Life Expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Not specified Renal: Glomerular filtration rate at least 50 mL/min Creatinine clearance at least 25 mL/min

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior systemic chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 1997-12; Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Harper, MD, Study Chair — St. Thomas' Hospital
Locations (62):
- Porto Alegre Hospital, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (4):
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
- Maria Hospital, Helsinki, Finland
- Antoni van Leeuwenhoekhuis, Amsterdam, Netherlands
- Christchurch Hospital, Christchurch, New Zealand
- Norwegian Radium Hospital, Oslo, Norway
- Groote Schuur Hospital, Cape Town, Cape Town, South Africa
- United Kingdom (52):
  - Royal United Hospital, Bath, England
  - University Birmingham, Birmingham, England
  - Children's Hospital - Birmingham UK, Birmingham, England
  - Bradford Hospitals NHS Trust, Bradford, England
  - Royal Sussex County Hospital, Brighton, England
  - Bristol Royal Hospital for Sick Children, Bristol, England
  - Bristol Oncology Centre, Bristol, England
  - Addenbrooke's NHS Trust, Cambridge, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Walsgrave Hospital, Coventry, England
  - Derbyshire Royal Infirmary, Derby, England
  - Derbyshire Children's Hospital, Derby, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Gloucester Royal NHS Trust - Glouchester Royal Hospital, Gloucester, England
  - Royal Surrey County Hospital, Guildford, England
  - Royal Free Hospital, Hampstead, London, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Cookridge Hospital, Leeds, England
  - St. James's Hospital, Leeds, England
  - University Hospitals of Leicester, Leicester, England
  - St. Bartholomew's Hospital, London, England
  - Guy's, King's and St. Thomas' Hospitals Trust, London, England
  - Westminster Hospital, London, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - University College Hospital, London, England
  - Manchester Children's Hospitals (NHS Trust), Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - South Tees Acute Hospitals NHS Trust, Middlesbrough, Cleveland, England
  - Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Hospital, Northwood, England
  - Norfolk & Norwich Hospital, Norwich, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Portsmouth Hospitals NHS Trust, Portsmouth, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Weston Park Hospital, Sheffield, England
  - Royal South Hants Hospital, Southampton, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden Hospital, Sutton, England
  - Princess Royal Hospital, Telford, England
  - Walsall Manor Hospital, Walsall, England
  - Southend General Hospital, Westcliff-on-Sea, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - Royal Infirmary, Glasgow, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Llandough Hospital, Penarth, Wales
  - Royal Preston Hospital, Preston

REFERENCES:
- [Result] Highley MS, Griffiths GO, Uscinska BM, Huddart RA, Barber JB, Parmar MK, Harper PG; NCRI Bladder Cancer Clinical Studies Group. A phase II trial of continuous 5-fluorouracil in recurrent or metastatic transitional cell carcinoma of the urinary tract. Clin Oncol (R Coll Radiol). 2009 Jun;21(5):394-400. doi: 10.1016/j.clon.2009.01.011. Epub 2009 Mar 9. PMID 19269798
- [Result] Highly M, Griffiths G, Uscinska B, et al.: A phase II trial of continous 5-fluorouracil (5-FU) in recurrent locally advanced or metastatic transitional cell of the urinary tract. Br J Cancer 85(suppl 1): A-P77, 52, 2001.